CLINICAL TRIAL: NCT06479460
Title: Director, Department of Pathology, Jiangsu Provincial People's Hospital
Brief Title: Clinical Application of ctDNA Dynamic Monitoring in Neoadjuvant Therapy for HER2-positive Breast Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: ClINICALRESEARCH-001
Record Dates: First submitted 2024-06-24; First posted 2024-06-28 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer; Neoadjuvant; HER2-positive Breast Cancer; Circulating Tumor DNA
Keywords: breast cancer; circulating tumor DNA; MRD
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collect peripheral blood samples from subjects at different treatment nodes, extract and test ctDNA nucleic acid samples for testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ctDNA-MRD — This study is an observational non intervention study that only tests peripheral blood samples from different treatment nodes of the subjects, without interfering with the normal clinical diagnosis and treatment process of the patients.

SUMMARY:
1. To explore the predictive value of ctDNA in HER2 positive breast cancer neoadjuvant therapy population;
2. To evaluate the prognostic value of ctDNA in HER2 positive breast cancer neoadjuvant therapy population.

DETAILED DESCRIPTION:
This study plans to enroll 50 HER2 positive breast cancer patients in early stage (T2-3, N0-1, M0)/local late stage (T2-3, N2-3, M0 or T4a-c, Nany, M0), collect baseline tumor tissue samples of patients, as well as peripheral blood samples of multiple nodes at baseline, during new adjuvant therapy, after new adjuvant therapy (before surgery), and after surgery, detect the mutation of tumor tissue through 1021 panel, and conduct ctDNA detection of peripheral blood samples based on personalized panel design based on tumor tissue specific mutations, to explore the efficacy prediction and prognostic predictive value of ctDNA in HER2 positive new adjuvant therapy population.

ELIGIBILITY:
Inclusion Criteria:

1. Women with breast cancer diagnosed clinically and pathologically, aged 18-75 years;
2. ECOG performance score is 0-1;
3. Histologically confirmed as early or locally advanced invasive breast cancer: the diameter of the primary tumor is more than 2 cm, and HER2 is positive (confirmed by IHC or FISH).
4. The patient did not receive any treatment for breast cancer before enrollment;
5. Having lesions measurable according to RECIST 1.1 standards;
6. The subjects voluntarily joined this study, signed an informed consent form, had good compliance, and cooperated with follow-up; 7) Breast cancer patients who plan to use neoadjuvant therapy.

Exclusion criteria

1. Patients with known metastatic or stage IV breast cancer;
2. There are other untreated malignant tumors other than breast cancer;
3. Patients with one or more serious systemic diseases that, in the eyes of researchers, can impair their ability to complete research;
4. According to the researchers' assessment, there may be other factors that could force the subjects to terminate the study midway, such as suffering from other serious illnesses (including mental illnesses) that require concurrent treatment, severe abnormal laboratory test values, family or social factors, which may affect the safety of the subjects or the collection of experimental data.
5. Unable to follow up with the study according to the determined clinical follow-up period;
6. Cannot accept or provide specified efficacy evaluation methods such as CT.
7. Unable to obtain sufficient tumor tissue samples or peripheral blood samples.

Exclusion Criteria:

- 1) Patients with known metastatic or stage IV breast cancer; 2) There are other incurable malignant tumors present; 3) One or more serious systemic diseases that, in the eyes of researchers, can impair the patient's ability to complete the study; 4) According to the researcher's judgment, there are other factors that may cause the subject to be forced to terminate the study midway, such as other serious illnesses (including mental illness) requiring concurrent treatment, severe abnormal laboratory test values, family or social factors, which may affect the safety of the subject or the collection of trial data.

5) Unable to follow the determined clinical follow-up period in conjunction with the study for follow-up; 6) Unable to accept or provide specified efficacy evaluation methods such as CT.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study plans to enroll 50 women patients with HER2 positive early (T2-3, N0-1, M0)/local late (T2-3, N2-3, M0 or T4a-c, Nany, M0) breast cancer, who can accept new adjuvant treatment, voluntarily sign the informed consent form, timely and sufficiently obtain tumor tissue and peripheral blood samples for testing, and are willing to cooperate with follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-03-08 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative pathological pCR rate | 2024.3 -- 2026. 3
  Postoperative pathological pCR rate of HER-2 positive breast cancer patients after completing neoadjuvant therapy and undergoing surgical resection

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Province Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Heitzer E, Haque IS, Roberts CES, Speicher MR. Current and future perspectives of liquid biopsies in genomics-driven oncology. Nat Rev Genet. 2019 Feb;20(2):71-88. doi: 10.1038/s41576-018-0071-5. PMID 30410101
- [Background] McDonald BR, Contente-Cuomo T, Sammut SJ, Odenheimer-Bergman A, Ernst B, Perdigones N, Chin SF, Farooq M, Mejia R, Cronin PA, Anderson KS, Kosiorek HE, Northfelt DW, McCullough AE, Patel BK, Weitzel JN, Slavin TP, Caldas C, Pockaj BA, Murtaza M. Personalized circulating tumor DNA analysis to detect residual disease after neoadjuvant therapy in breast cancer. Sci Transl Med. 2019 Aug 7;11(504):eaax7392. doi: 10.1126/scitranslmed.aax7392. PMID 31391323
- [Background] Rothe F, Silva MJ, Venet D, Campbell C, Bradburry I, Rouas G, de Azambuja E, Maetens M, Fumagalli D, Rodrik-Outmezguine V, Di Cosimo S, Rosa D, Chia S, Wardley A, Ueno T, Janni W, Huober J, Baselga J, Piccart M, Loi S, Sotiriou C, Dawson SJ, Ignatiadis M. Circulating Tumor DNA in HER2-Amplified Breast Cancer: A Translational Research Substudy of the NeoALTTO Phase III Trial. Clin Cancer Res. 2019 Jun 15;25(12):3581-3588. doi: 10.1158/1078-0432.CCR-18-2521. Epub 2019 Mar 12. PMID 30862692
- [Background] Cailleux F, Agostinetto E, Lambertini M, Rothe F, Wu HT, Balcioglu M, Kalashnikova E, Vincent D, Viglietti G, Gombos A, Papagiannis A, Veys I, Awada A, Sethi H, Aleshin A, Larsimont D, Sotiriou C, Venet D, Ignatiadis M. Circulating Tumor DNA After Neoadjuvant Chemotherapy in Breast Cancer Is Associated With Disease Relapse. JCO Precis Oncol. 2022 Sep;6:e2200148. doi: 10.1200/PO.22.00148. PMID 36170624
- [Background] Magbanua MJM, Swigart LB, Wu HT, Hirst GL, Yau C, Wolf DM, Tin A, Salari R, Shchegrova S, Pawar H, Delson AL, DeMichele A, Liu MC, Chien AJ, Tripathy D, Asare S, Lin CJ, Billings P, Aleshin A, Sethi H, Louie M, Zimmermann B, Esserman LJ, van 't Veer LJ. Circulating tumor DNA in neoadjuvant-treated breast cancer reflects response and survival. Ann Oncol. 2021 Feb;32(2):229-239. doi: 10.1016/j.annonc.2020.11.007. Epub 2020 Nov 21. PMID 33232761